CLINICAL TRIAL: NCT03196193
Title: Randomized Controlled Study Comparing Zimmer Natural Nail System Cephalomedullary Asia Nail With Anterior Support Screw (AS2) Versus Conventional Technique
Brief Title: CM Asia Nail With AS2 Without AS2 （AS2 Study）
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T.CR.I.AP.16.4
Record Dates: First submitted 2017-03-28; First posted 2017-06-22 (Actual); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Trochanteric Fracture of Femur
MeSH Terms: interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Intervention Model Description: At surgery, intervention group using ZNN CM Asia with AS2 technique. At surgery, conventional group using ZNN CM Asia without AS2 technique.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: (Investigational group) or ZNN CM Asia without AS2 technique (Control group). The randomization scheme is based on equal numbers per group. The randomization will occur via a random number generator (computer) using a blocked randomization procedure. The block size will not be disclosed to the sites, and the doctor or other health care professional will not have influence on the randomization scheme. Sealed opaque envelopes, which will be prepared based on predetermined randomization assignment, will be provided to each study site before study initiation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ZNN CM Asia with AS2 technique (Experimental): Open Reduction and Internal Fixation with AS2 Trochanteric Fracture treated by Open Reduction and Internal Fixation using with ZNN CM Asia nail.
  Bone fragment will be stabilized by additional screw fixation (Anterior Support Screw).
  Interventions: Procedure: Open Reduction and Internal Fixation; Device: ZNN CM Asia; Device: Anterior Support Screw
- ZNN CM Asia without AS2 technique (Active Comparator): Trochanteric Fracture treated by Open Reduction and Internal Fixation using with ZNN CM Asia nail without additional screw fixation.
  Interventions: Procedure: Open Reduction and Internal Fixation; Device: ZNN CM Asia

INTERVENTIONS:
Procedure: Open Reduction and Internal Fixation — Fractured bone fragments are reduced and stabilized by intramedullary nail.
Device: ZNN CM Asia — Reduced bone fragments are to be stabilized by Zimmer Natural Nail CM Asia System.
Device: Anterior Support Screw — Experimental group will receive insertion of ACE 4.5/5.0mm cannulated lag-screw anteriorly to Zimmer Natural Nail CM Asia Lag-screw.
  Other Names: ACE 4.5/5.0mm cannulated lag-screw
  Arms: ZNN CM Asia with AS2 technique

SUMMARY:
The purpose of this study is to compare reduction positon maintenance rate at 3 weeks post-operatively between patients operated with Anterior Support Screw (AS2) and without AS2 technique in RCT setting. Total 240 cases(each arm 120 cases) will be enrolled at maximum 15sites, total study duration is 22months.

DETAILED DESCRIPTION:
Objective： To compare fracture reduction maintenance rate at 2-3weeks post-operatively between patients operated with AS2 (investigational group) and patients operated without AS2 (Control group) using same implant system (ZNN CM Asia, Zimmer Biomet).

Endpoint： Primary： The rate of reduction position maintenance at 2-3 weeks post-operatively. Secondary： Surgery time / fracture type / postoperative reduction position / CT assessment / Safety information

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria.

* Eligible for intramedullary nailing.
* Fracture type is classified as 3-partB or 4-part fracture in 3D-CT (Three Dimensional Computed Tomography) classification (Nakano), and combination with a subtype P in lateral classification (Ikuta) at preoperative CT (Computed Tomography) assessment.(In the case of classified in radiograph (X-ray) at preoperative: Classified as Type 4 or Type 5 in Jensen classification, and combination of subtype P in lateral classification (Ikuta))
* Japanese Male or female
* > 20 years of age
* Primary closed intertrochanteric fracture of the femur
* Subjects willing to return for follow-up evaluations.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study.

* Patient who cannot take CT image within 3 days and 2-3weeks after surgery.
* Uncooperative patient or patient with neurologic disorders who are incapable of following directions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Maehara, MD, Ph. D, Principal Investigator — Kagawa Rosai Hospital
Locations (12):
- Japan (12):
  - Kure Kyosai Hospital, Kure, Hiroshima
  - Toyooka Hospital, Toyooka, Hyōgo
  - Kasugai Municipal Hospital, Aichi, Kasugai
  - Hoshigaoka Medical Center, Hirakata, Osaka
  - Numazu City Hospital, Numazu, Shizuoka
  - Saiseikai Takaoka Hospital, Takaoka, Toyama
  - Kyushu Central Hospital, Fukuoka
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Niigata Central Hospital, Niigata
  - Okayama Red Cross Hospital, Okayama
  - Okayama Rosai Hospital, Okayama
  - Saga Pref. Medical Centre Koseikan, Saga

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ZNN CM Asia With AS2 Technique: Open Reduction and Internal Fixation with AS2 Trochanteric Fracture treated by Open Reduction and Internal Fixation using with ZNN CM Asia nail.
  Bone fragment will be stabilized by additional screw fixation (Anterior Support Screw).
  Open Reduction and Internal Fixation: Fractured bone fragments are reduced and stabilized by intramedullary nail.
  ZNN CM Asia: Reduced bone fragments are to be stabilized by Zimmer Natural Nail CM Asia System.
  Anterior Support Screw: Experimental group will receive insertion of ACE 4.5/5.0mm cannulated lag-screw anteriorly to Zimmer Natural Nail CM Asia Lag-screw.
Period: Overall Study
Arm/Group | ZNN CM Asia With AS2 Technique | ZNN CM Asia Without AS2 Technique
Started | 121 | 119
Completed | 118 | 119
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Computed Tomography (CT) data missing | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZNN CM Asia With AS2 Technique | ZNN CM Asia Without AS2 Technique | Total
Number analyzed (Participants) | 118 | 119 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 85.9 (8.9) | 86.7 (7.9) | 86.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 97 | 200
  Male | 15 | 22 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 118 | 119 | 237
Height [Mean (Standard Deviation); unit: cm] | 148.9 (8.8) | 150.0 (9.0) | 149.4 (8.9)
Weight [Mean (Standard Deviation); unit: kg] | 45.3 (9.8) | 46.2 (9.3) | 45.8 (9.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patient With and Without Excessive Lag Screw Sliding Distance
Description: Number of patient was counted based on CT measurement results. Relative position of lag screw between CT images taken at both immediate and 2-3 weeks postoperatively was measured and recorded in value (e.g., 1.5 mm). This was called as "lag screw sliding distance". Four millimeter was set as threshold to define success and failure. Less than 4mm of lag screw sliding distance was recognized as Success and equal to or more than 4mm of lag screw sliding distance was recognized as Failure.
Time Frame: Postoperative 2-3 week
Measure: Count of Participants; unit: Participants
Arm/Group | ZNN CM Asia With AS2 Technique | ZNN CM Asia Without AS2 Technique
Number analyzed (Participants) | 118 | 119
Participants
  Success (lag screw sliding distance <4mm) | 109 | 97
  Failure (lag screw sliding distance >=4mm) | 9 | 22

2. Secondary Outcome: Surgery Time
Description: Surgery time from skin incision to closure
Time Frame: Intraoperative, an average of 1 hour
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ZNN CM Asia With AS2 Technique | ZNN CM Asia Without AS2 Technique
Number analyzed (Participants) | 118 | 119
minutes | 68.2 (21.8) | 59.8 (20.9)

3. Secondary Outcome: Image Assessment Using Computed Tomography (CT)
Description: Number of patient was counted based on CT measurement results. When the fracture reduction position achieved at surgery was maintained at 2 to 3 weeks, then the patient was categorized as success (Reduction position maintained). On the other hand, patient was categorized as failure (Reduction position changed) in the case that the fracture reduction position was changed.
  Fracture repair position was categorized into three; "Anterior", "Neutral" or "Posterior" based on relative position of proximal bone fragment and distal bone fragment.
  This analysis only includes patients whose fracture reduction position at immediate postoperative CT was either "Anterior" or "Neutral".
  If both immediate and 2-3 weeks postoperative CT images show same fracture reduction position (example: "Anterior" at immediate postoperatively & "Anterior" at 2-3 weeks postoperatively), then the patient was recognized as Success (Reduction position maintained).
Time Frame: 2-3 weeks postoperatively
Population: Participants, whose immediate postoperative reduction position is assessed as either "Anterior" or "Neutral", were eligible.
  Eight patients in ZNN CM Asia with AS2 technique group and 6 patients in ZNN CM Asia without AS2 technique group were excluded from this analysis (their immediate postoperative reduction position was "Posterior".)
Measure: Count of Participants; unit: Participants
Arm/Group | ZNN CM Asia With AS2 Technique | ZNN CM Asia Without AS2 Technique
Number analyzed (Participants) | 110 | 113
Participants
  Reduction position maintained | 104 | 92
  Reduction position changed | 6 | 21

4. Secondary Outcome: Intraoperative Safety
Description: This is to evaluate whether any adverse events specific to insert additional screw for AS2 technique were occurred.
Time Frame: Intraoperative
Population: Intent-to-treat group
Measure: Count of Participants; unit: Participants
Arm/Group | ZNN CM Asia With AS2 Technique | ZNN CM Asia Without AS2 Technique
Number analyzed (Participants) | 121 | 119
Participants
  No adverse event | 121 | 119
  adverse event | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 weeks after surgery
Arm/Group | ZNN CM Asia With AS2 Technique | ZNN CM Asia Without AS2 Technique
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/119
Serious Adverse Events (participants affected / at risk) | 1/121 | 0/119
Other Adverse Events (participants affected / at risk) | 0/121 | 0/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZNN CM Asia With AS2 Technique (N=121) | ZNN CM Asia Without AS2 Technique (N=119)
Cut-out (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Proximal fracture fragment was dislodged after surgery and required reoperation to hemi hip replacement surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT03196193/Prot_SAP_000.pdf